CLINICAL TRIAL: NCT03832894
Title: Effects of Adding Oestradiol Supplementation in Luteal Phase in Patients Undergoing in Vitro Fertilization/ Intra Cytoplasmic Sperm Injection (IVF/ICSI ) Long Agonist Fresh Embryo Transfer Cycles
Brief Title: Oestradiol Supplementation in Luteal Long Agonist Fresh In Vitro Fertilization/Intra Cytoplasmic Sperm Injection ( IVF/ICSI) Cycle .
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, sherine Hosny Mohamed Gad Allah, Assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MD IVF
Record Dates: First submitted 2019-02-04; First posted 2019-02-06 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Infertility
Keywords: IVF; ICSI; oestradiol; long protocol
MeSH Terms: conditions — Infertility | interventions — Estradiol

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Randomization will be held by using the computer generated randomization codes, which will then be placed in the sealed envelopes by a third party (nurse).
  Each patient will choose a sealed envelope containing randomization number either group A or B. Both participant and health provider will be blinded to patients grouping
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group receiving oestradiol tablets in addition to progesterone (Active Comparator): Group A :Will receive 400mg progesterone in the form of vaginal or rectal suppositories in addition to estradiol valerate oral tablets in a dose of 4mg/day(2x2), for luteal phase support. Starting from the day of ovum pickup and for 14 days after embryo transfer.
  Group B : Will receive a dose of 400mg progesterone in the form of vaginal or rectal suppositories in addition to 2 placebo oral tablets(similar to estrogen tablets) for luteal phase support, from the day of Ovum pickup and for 14 days after embryo transfer.
  Interventions: Drug: Estradiol Valerate
- Group not receiving oestradiol tablets. (Placebo Comparator): Group B : Will receive a dose of 400mg progesterone in the form of vaginal or rectal suppositories in addition to 2 placebo oral tablets(similar to estrogen tablets) for luteal phase support, from the day of Ovum pickup and for 14 days after embryo transfer
  Interventions: Drug: Estradiol Valerate

INTERVENTIONS:
Drug: Estradiol Valerate — Oestradiol supplementation starting from day of trigger through out the luteal phase
  Other Names: Progynova; Progesterone vaginal suppositories

SUMMARY:
Whether oestradiol administration affects the pregnancy rate in long agonist fresh IVF/ICSI cycles. Oestradiol level will be measured the day of HCG trigger to assess whether oestradiol level affects cycle outcome results.

DETAILED DESCRIPTION:
6. Background and Rationale: Progesterone is essential for successful implantation and maintenance of early pregnancy . Although the oestrogen is not essential, it is important to maintain the progesterone level during the pregnancy and promote the transformation of the endometrium from the secretory to proliferative phase.

Compromised granulosa cells luteinisation could cause infertility or early miscarriage. In assisted reproductive technologies (ART) cycles, curettage of the granulosa cells during oocyte retrieval is thought to reduce corpora lutea function and thus progesterone production, resulting in a decrease in pregnancy rate.

Therefore, luteal support is routinely performed in ART cycles. Consensus has been reached on the supplementation of progesterone after the day of oocyte retrieval, which was performed in approximately 80% of the cycles and significantly improved clinical outcomes.However, the efficacy of oestradiol supplementation in luteal support remains controversial.

Previous studies have shown that the lower the serum estrogen level was at 4, 7 and 9 days following transplantation, the lower the clinical pregnancy rate. Previous studies showed that in patients with long or short duration ovulation induction, luteal support with oestradiol supplementation led to an increased serum estrogen level and an improved pregnancy rate . It was also found that patients having luteal support with estrogen (4 mg per day) had a significantly higher clinical pregnancy rate (40.6% vs 21.6%) and a significantly lower abortion rate (12.8% vs 38%) than those treated with progesterone alone.

In contrast, other investigators have failed to show any benefit of oestradiol supplementation during the luteal phase and a Cochrane review published in 2015 reported no differences in rates of live birth or ongoing pregnancy between the progesterone group and progesterone add oestrogen group. Hence, it remains unclear whether the addition of estrogen to progesterone for luteal support is associated with higher pregnancy rate and live birth rate.

In this study, the investigators will evaluate outcomes of patients undergoing IVF/ICSI-ET with oestradiol supplementation in addition to progesterone for luteal support. The investigators also report on the efficacy implications of oestradiol supplementation for patients undergoing IVF/ICSI-ET.

ELIGIBILITY:
Inclusion criteria:

1. Age group 20-38 years old.
2. Patients Undergoing gonadotropin Releasing Hormone (Gn RH) long agonist protocol, with fresh embryo transfer.
3. Day 3 Grade 1 embryos.
4. Trilamellar endometrium with ranging endometrial thickness from 8 mm to 14 mm.

Exclusion criteria:

1. Karyotypic abnormalities in either partner.
2. Patients with uterine abnormalities.
3. G3-G4 quality embryos.
4. Estradiol level 10,000 or more at time of trigger.
5. Cases of egg donation/sperm donation/embryo donation.
6. Polycystic ovary syndrome (PCOS )patients.
7. Poor responders (maternal age >40, Antral follicle counts (AFC )<5, Anti Mullerian Hormone (AMH )<1 and previous trial <5 oocyte retrieved ) (bologna criteria 2011)
8. Those with 3 or more implantation failure.
9. Endometrial thickness <8 or >14mm.
10. Severe male factor.

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Implantation rate | 4 weeks after embryo transfer of each enrolled patient
  Number of gestational sacs per number of embryos transferred per cycle

SECONDARY OUTCOMES:
Chemical pregnancy rate | Two weeks after embryo transfer of each enrolled patient
  Quantitative Beta Human Chorionic Gonadotropin (BHCG)
Clinical pregnancy rate | 4 weeks after embryo transfer of each enrolled patient with positive pregnancy test or 6 weeks from IVF cycle beginning in pregnant patients
  Intrauterine gestational sac with fetal pole with positive pulsation
Ongoing pregnancy rate | 10 weeks after embryo transfer of each enrolled patient or 12 weeks from starting IVF cycle in pregnant patients
  12 weeks gestation and more

CONTACTS AND LOCATIONS:
Locations (1):
- Art Unit/ Obatetrics and Gynecology Department, Cairo, Cair0, Egypt

IPD SHARING:
Plan to Share IPD: Undecided